CLINICAL TRIAL: NCT01651299
Title: Observational Study of Recovery From Copperhead Snake Envenomation
Brief Title: Copperhead Envenomation Observational Study
Status: Completed | Type: Observational
Sponsor: BTG International Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: BTG-PR005-001
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2012-09

CONDITIONS: Copperhead Snake Envenomation
Keywords: copperhead snake envenomation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of the study is to evaluate the responsiveness and utility of several clinical outcome assessments in the setting of copperhead snakebite. The secondary objective is to characterize the clinical course of signs, symptoms and impairment during the recovery phase of copperhead snakebite.

DETAILED DESCRIPTION:
This observational study will document the patient's recovery from copperhead snakebite. All care provided will be at the discretion of the treating physician in accordance with the local standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Envenomation by a copperhead snake
* Presentation for care at a health care facility within 24 hrs of envenomation
* Envenomation on an extremity distal to the knee or elbow
* Clinical evidence of venom effect (limb swelling and/or tenderness)
* Enrollment can be completed within 48 hrs of envenomation prior to discharge
* Patient is willing and able to complete follow-up schedule of assessments
* Patient is able to read, comprehend and sign IRB approved informed consent
* Patient is able to read and comprehend written assessment tools
* Patient is at least 18 yrs old
* Patient is sober, competent and able to complete verbal and written informed consent

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is a prisoner
* Patient has distracting injury, condition with acute pain or functional impairment, and/or is unable to make a reliable self-report of status
* Patient has had previous snake envenomation to any body area within 30 days prior to screening/enrollment, regardless of whether antivenom was administered
* Patient had an acute traumatic or medical event, surgery, or exacerbation of pre-existing medical or surgical condition effecting the envenomated extremity within 30 days prior to screening/enrollment
* Patient has participated in a clinical study involving and investigational pharmaceutical product or device within 3 months prior to screening that may have impact on clinical outcomes of snakebite
* Patient has previously participated in this study
* Patient is, in the investigator's opinion, otherwise unsuitable for participation. Note: Treatment with antivenom prior to eligibility evaluation is not an exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and non-pregnant females at least 18 yrs of age with evidence of copperhead envenomation on an extremity distal to the knee or elbow that present for care at a health care facility within 24 hours of envenomation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Patient Global Assessment of Recovery (PGAR) | Time of Discharge, Day 3, Day 7, Day 14, Day 21, and Day 28
Numeric Pain Rating Scale (NPRS) | Time of Discharge, Day 3, Day 7, Day 14, Day 21, and Day 28
Numeric Swelling Score (NSS) | Time of Discharge, Day 3, Day 7, Day 14, Day 21, and Day 28
SF36v2 (Acute Version) | Time of Discharge, Day 7, Day, 14, Day 21, and Day 28
Swelling Figure-of-8 Measurement | Time of Discharge, Day 3, Day 7, Day 14, Day 21, and Day 28
Grip Strength | Time of Discharge, Day 3, Day 7, Day 14, Day 21, and Day 28
Walking Speed | Time of Discharge, Day 3, Day 7, Day 14, Day 21, and Day 28
Patient Global Impression of Change (PGIC) | Time of Discharge, Day 3, Day 7, Day 14, Day 21, and Day 28
Return to Work/School/ADLs | Day 3, Day 7, Day 14, Day 21, and Day 28
Patient-Specific Functional Scale (PSFS) | Day 3, Day 7, Day 14, Day 21, and Day 28
WPAI:SHP V2 | Day 3, Day 7, Day 14, Day 21, and Day 28
Disorders of the Arm, Shoulder, and Hand (DASH) | Time of Discharge, Day 3, Day 7, Day 14, Day 21, and Day 28
Lower Extremity Functional Scale | Time of Discharge, Day 3, Day 7, Day 14, Day 21, and Day 28

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - LSU Health Sciences Center, Shreveport, Louisiana
  - University of Mississippi Medical Center, Jackson, Michigan
  - Washington University, St Louis, Missouri
  - Duke Medical Center, Durham, North Carolina
  - Vidant Health, Greenville, North Carolina
  - St. Joseph Regional Health Center, Bryan, Texas
  - Harris Methodist Hospital, Fort Worth, Texas
  - Scott and White Hospital, Temple, Texas
  - University of Virginia, Blue Ridge PC, Charlottesville, Virginia
  - Virginia Commonwealth University Richmond, Richmond, Virginia

REFERENCES:
- [Derived] Lavonas EJ, Gerardo CJ; Copperhead Snakebite Recovery Outcome Group. Prospective study of recovery from copperhead snake envenomation: an observational study. BMC Emerg Med. 2015 May 15;15:9. doi: 10.1186/s12873-015-0033-6. PMID 25975429